CLINICAL TRIAL: NCT05135559
Title: Open-label Study Investigating Efficacy, Safety and Pharmacokinetics of Concizumab Prophylaxis in Children Below 12 Years With Haemophilia A or B With or Without Inhibitors
Brief Title: A Research Study on How Well Concizumab Works for You if You Have Haemophilia A or B With or Without Inhibitors
Acronym: Explorer10
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7415-4616; U1111-1247-7330 (Other: World Health Organization (WHO)); 2020-000504-11 (EudraCT Number); jRCT2031220097 (Registry Identifier: JAPIC)
Expanded Access: NCT04921956 (Available)
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A and B With and Without Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — concizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Concizumab-naïve patients (Experimental): Concizumab-naïve participants below 12 years of age at the time of consent/assent
  Interventions: Drug: Concizumab
- Patients coming from compassionate use (Experimental): Patients previously treated with concizumab via compassionate use, either on an individual patient basis or through the concizumab compassionate use programme NN7415-4807
  Interventions: Drug: Concizumab

INTERVENTIONS:
Drug: Concizumab — Participants in Arm 1 will be assigned to concizumab prophylaxis starting with a loading dose on treatment day 0 followed by daily injections of an individual maintenance dose.
  Participants in Arm 2 will be assigned to concizumab prophylaxis with daily injections of an individual maintenance dose.

SUMMARY:
This study will test how well a new medicine called concizumab works for participants who have haemophilia A or B with or without inhibitors. The purpose is to show that concizumab can prevent bleeds and is safe to use.

Participants will have to inject the study medicine every day under the skin with a pen-injector.

The study will last for at least 2 years and up to about 4 years. The length of time the participant will be in the study depends on if the study medicine will be available for purchase in their country.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Diagnosis of congenital severe haemophilia A (FVIII below 1%) or moderate/severe congenital haemophilia B (FIX (coagulation factor IX) below or equal to 2%), or congenital haemophilia with inhibitors.
* For arm 1 only: Male aged below 12 years of age at the time of signing informed consent.
* For arm 1 only: Patients with inhibitors (haemophilia A with inhibitors or haemophilia B with inhibitors)

  1. Patients with HAwI (haemophilia A with inhibitors) with historical medical records of a total of at least 26 weeks of on-demand treatment (On-demand or PPX treatment qualifying for this study is understood as patient-treatment solely for bleeds with intravenous coagulation factor-containing products) within the last 52 weeks prior to enrolment (For patients below 1 year of age that have been diagnosed with haemophilia <1 year prior to enrolment, historical medical records from time of diagnosis will suffice as long as medical records of a total of at least 26 weeks of relevant treatment is available).
  2. Patients with HBwI (haemophilia B with inhibitors) with historical medical records of a total of at least 26 weeks of on-demand treatment (On-demand or PPX treatment qualifying for this study is understood as patient-treatment solely for bleeds with intravenous coagulation factor-containing products) within the last 52 weeks prior to enrolment (For patients below 1 year of age that have been diagnosed with haemophilia <1 year prior to enrolment, historical medical records from time of diagnosis will suffice as long as medical records of a total of at least 26 weeks of relevant treatment is available).
  3. Patients with HBwI regardless of the regimen and duration of previous haemophilia treatment (On-demand or PPX treatment qualifying for this study is understood as patient-treatment solely for bleeds with intravenous coagulation factor-containing products)
* For arm 1 only: Patients without inhibitors (haemophilia A or haemophilia B)

  1. Patients with historical medical records of at least 52 weeks of on-demand treatment (On-demand or PPX treatment qualifying for this study is understood as patient-treatment solely for bleeds with intravenous coagulation factor-containing products; Surgery related PPX or short-term PPX (e.g., in relation to a severe bleed) is not allowed) during the last year prior to enrolment and with at least 3 documented treated bleeds (For participants less than (<) 2 years of age there is no limitation for number of documented treated bleeds in the medical history) during this period
  2. Patients with historical medical records of a total of at least 26 weeks of PPX (prophylaxis) treatment (On-demand or PPX treatment qualifying for this study is understood as patient-treatment solely for bleeds with intravenous coagulation factor-containing products) within the last 52 weeks prior to enrolment (For patients below 1 year of age that have been diagnosed with haemophilia <1 year prior to enrolment, historical medical records from time of diagnosis will suffice as long as medical records of a total of at least 26 weeks of relevant treatment is available)
* For arm 2 only: Male patients (regardless of age) previously treated with concizumab via compassionate use.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention or related products.
* Known inherited or acquired coagulation disorder other than congenital haemophilia.
* Ongoing or planned Immune Tolerance Induction treatment.
* History of thromboembolic disease (aIncludes arterial and venous thrombosis including myocardial infarction, pulmonary embolism, cerebral infarction/thrombosis, deep vein thrombosis, other clinically significant thromboembolic events and peripheral artery occlusion.). Current clinical signs of or treatment for thromboembolic disease. Patients who in the judgement of the investigator are considered at high risk of thromboembolic events (Thromboembolic risk factors could include, but are not limited to, hypercholesterolemia, diabetes mellitus, hypertension, obesity, smoking, family history of thromboembolic events, arteriosclerosis, other conditions associated with increased risk of thromboembolic events).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2026-04-21 (Estimated); Study Completion 2029-11-02 (Estimated)

PRIMARY OUTCOMES:
For inhibitor patients with at least 26 weeks on-demand treatment during the last 52 weeks prior enrolment: Number of treated spontaneous and traumatic bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients treated on demand during at least the last 52 weeks prior enrolment: Number of treated spontaneous and traumatic bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)

SECONDARY OUTCOMES:
For inhibitor patients with at least 26 weeks on-demand treatment during the last 52 weeks prior enrolment: Number of all bleeding episodes (spontaneous and traumatic) | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For inhibitor patients with at least 26 weeks on-demand treatment during the last 52 weeks prior enrolment: Number of treated spontaneous bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For inhibitor patients with at least 26 weeks on-demand treatment during the last 52 weeks prior enrolment: Number of treated joint bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For inhibitor patients with at least 26 weeks on-demand treatment during the last 52 weeks prior enrolment: Number of treated bleeding episodes in baseline target joints | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients treated on-demand during at least the last 52 weeks prior enrolment: Number of all bleeding episodes (spontaneous and traumatic) | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients treated on-demand during at least the last 52 weeks prior enrolment: Number of treated spontaneous bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients treated on-demand at least the last 52 weeks prior enrolment: Number of treated joint bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients treated on-demand at least the last 52 weeks prior enrolment: Number of treated bleeding episodes in baseline target joints | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients with at least 26 weeks PPX treatment during the last 52 weeks prior enrolment: Number of treated spontaneous and traumatic bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients with at least 26 weeks PPX treatment during the last 52 weeks prior enrolment: Number of all bleeding episodes (spontaneous and traumatic) | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients with at least 26 weeks PPX treatment during the last 52 weeks prior enrolment: Number of treated spontaneous bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients with at least 26 weeks PPX treatment during the last 52 weeks prior enrolment: Number of treated joint bleeding episodes | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
For non-inhibitor patients with at least 26 weeks PPX treatment during the last 52 weeks prior enrolment: Number of treated bleeding episodes in baseline target joints | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of episode(s)
Concizumab-naïve pateints - Number of treatment emergent adverse events, reported both separately for inhibitor and non-inhibitor patients and combined | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of event(s)
Number of thromboembolic events, reported both separately for inhibitor and non-inhibitor patients and combined | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of event(s)
Number of hypersensitivity type reactions, reported both separately for inhibitor and non-inhibitor patients and combined | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of event(s)
Number of injection site reactions, reported both separately for inhibitor and non-inhibitor patients and combined | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of event(s)
Number of patients who develop antibodies to concizumab - yes/no, reported both separately for inhibitor and non-inhibitor patients and combined | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of patient(s)
Number of treatment emergent adverse events, reported both separately for inhibitor and non-inhibitor patients and combined | From start of treatment (week 0) up until the primary analysis cut-off (at least 32 weeks)
  Count of event(s)
Concizumab plasma concentrations prior to dosing, reported both separately for inhibitor and non-inhibitor patients and combined | Week 32
  Measured in ng/mL
Peak thrombin generation prior to dosing, reported both separately for inhibitor and non-inhibitor patients and combined | Week 32
  Measured in nM
Free TFPI concentration prior to dosing, reported both separately for inhibitor and non-inhibitor patients and combined | Week 32
  Measured in ng/mL
Pre-dose (trough) concizumab plasma concentration (Ctrough), reported both separately for inhibitor and non-inhibitor patients and combined | Prior to the concizumab administration at week 20
  Measured in ng/mL
Maximum concizumab plasma concentration (Cmax), reported both separately for inhibitor and non-inhibitor patients and combined | From 0 to 24 hours where 0 is the time of the concizumab dose at week 20
  Measured in ng/mL
Area under the concizumab plasma concentration-time curve (AUC), reported both separately for inhibitor and non-inhibitor patients and combined | From 0 to 24 hours where 0 is the time of the concizumab dose at week 20
  Measured in ng*hr/mL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (90):
- United States (19):
  - Rady Childrens Hosp San Diego, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Arnold Palmer Children's Hospital, Orlando, Florida
  - Nemours Child Orlando Hem/Onc., Orlando, Florida
  - Augusta Univ/Childrens Hosp-GA, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Childrens Hospital of Chicago, Chicago, Illinois
  - Indiana Hemophilia-Thromb Ctr, Indianapolis, Indiana
  - Children's Hosp-New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Children's Nebraska, Omaha, Nebraska
  - ECU Sickle Cell Comp Clinic, Greenville, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - St Christopher Hosp for Child, Philadelphia, Pennsylvania
  - Vanderbilt Hemostasis Treatment Clinic, Nashville, Tennessee
  - Cook Children's Hospital-Hematology-Oncology, Fort Worth, Texas
  - Texas Children's Hospital_Houston, Houston, Texas
  - Pediatrics Hematology/Oncology Clinic Battle Building, Charlottesville, Virginia
- Algeria (2):
  - Haematology and Blood Bank Department, Algiers
  - CHU Constantine BEN BADIS/ Hematology department, Constantine
- Bosnia and Herzegovina (2):
  - University Clinical Center of Republic Srpska (545), Banja Luka
  - University Clinical Centre Tuzla, Tuzla
- Bulgaria (3):
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Pediatrics, Plovdiv
  - UMHAT Tsaritsa Yoanna - ISUL EAD, Pediatric clinical hematology and oncology, Sofia
  - UMHAT "Sveta Marina" EAD, Varna
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
- Tallinn Children's Hospital, Tallinn, Estonia
- France (3):
  - Centre Hospitalier Metropole Savoie, Chambéry
  - Ap-Hp-Hopital de Bicetre-1, Le Kremlin-Bicêtre
  - AP-HP-HOPITAL NECKER_Service d'hématologie, Paris
- Greece (2):
  - Aghia Sophia Childrens' Hospital, Athens
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
- India (11):
  - Guwahati Medical College, Guwahati, Assam
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - SSSH_Dept. of Clinical Haematology & Haemato Oncology, Kolhāpur, Maharashtra
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - K.J Somaiya Hospital and Research Centre, Mumbai, Maharashtra
  - MCGM - Comprehensive Thalassemia Care, Mumbai, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - S.C.B. Medical College, Cuttack, Odisha
  - J K Lon Hospital, Jaipur, Rajasthan
  - Post Graduate Institute of Child Health, Noida, Uttar Pradesh
  - SGPGI, Lucknow, Uttart Pradesh
- Italy (4):
  - A.O.U policlinico "G. Rodolico-San Marco", Catania
  - Dipartimento di Ematologia Univ. Firenze, Florence
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera-Universitaria Parma, Parma
- Japan (2):
  - St. Marianna University School of Medicine Hospital_Pediatrics, Kanagawa
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
- Lebanon (2):
  - Saint George Hospital University Medical Center, Beirut
  - Hospital Nini, Tripoli
- Centre of Oncology and Hematology, Vilnius University, Vilnius, Lithuania
- Malaysia (4):
  - Hospital Tunku Azizah, Kampung Baru, Kuala Lumpur
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu
- PHI University Clinic for Children's Diseases Skopje, Skopje, North Macedonia
- Klinisk forskningspost, Oslo, Norway
- Poland (4):
  - Uniwersytecki Szpital Kliniczny im. J.Mikulicza-Radeckiego, Wroclaw, Lower Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dzieciecy, Dzial Krwiolecznictwa, Lublin
  - Uniwersyteckie Centrum Kliniczne WUM, Warsaw
- Romania (3):
  - Clinic of Haematology, Fundeni Clinical Institute, Bucharest
  - Spitalul Clinic de Urgenta pentru Copii Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean De Urgenta Bihor, Oradea
- Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng, South Africa
- Spain (4):
  - Hospital Virgen de la Arrixaca - Hematología, El Palmar, Murcia
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- Koagulationscentrum, Gothenburg, Sweden
- Thailand (5):
  - Sunpasitthiprasong Hospital_Pediatrics Department, Ubon Ratchathani, Mueang Distirct,
  - King Chulalongkorn Memorial Hospital_Bangkok_0, Bangkok
  - King Chulalongkorn Memorial Hospital_Pediatric Hematology-Oncology, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital - Hematology and Oncology, Bangkok
- Turkey (Türkiye) (8):
  - Gazi University, Ankara, Beşevler/Ankara
  - Gazi Üniversitesi Hastanesi- Hematoloji, Ankara, Beşevler/Ankara
  - Acibadem Adana Hastanesi, Adana
  - Acıbadem Adana Hastanesi-Hematoloji, Adana
  - Ege Universitesi Tip Fakultesi, Izmir
  - Ege Üniversitesi Hastanesi- Hematoloji, Izmir
  - Ondokuz Mayis University Medical Faculty Ped. Haematology, Samsun
  - Ondokuz Mayıs Üniversitesi Hastanesi - Hematoloji, Samsun
- United Kingdom (4):
  - Birmingham Children's Hospital, Birmingham
  - University Hospitals Bristol & Weston NHS Foundation Trust, Bristol
  - Evelina London Children's Hospital - Haemophilia, London
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com